CLINICAL TRIAL: NCT02204189
Title: The Clinical Study of Acute Pancreatitis With Gastrointestinal Dysfunction Treated by TongFuSan for External Application on ShenQue Acupoint
Brief Title: The Clinical Study of Acute Pancreatitis Treated by TongFuSan
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, miaobin, associate chief physician, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: z141100002114004
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis; gastrointestinal dysfunction; TongFuSan; ShenQue acupoint
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TongFuSan (Experimental): TongFuSan 1g per time, change every day, the duration is seven days
  Interventions: Drug: TongFuSan

INTERVENTIONS:
Drug: TongFuSan — TongFuSan 1g

SUMMARY:
The purpose of this study is to determine whether TongFuSan is effective in the treatment of acute pancreatitis with gastrointestinal dysfunction.

DETAILED DESCRIPTION:
* Patient who is diagnosed with acute pancreatitis(AP) should be included.
* Patients will be divided into two groups as random number table: control group(A) and experimental group(B).
* Group A will be given Mosapride po,and group B will be given TongFusan except for basic treatments of AP.
* Same investigator will write the case report form.
* Investigator will collect the patients' blood in three points: on admission, the third day and the seventh day.
* Otherwise, we need write down patients' clinical manifestation,Traditional Chinese Medicine differentiation, the result of clinical tests.
* When the patient discharge, we will write down the treatment measures, therapeutic effect, length of stay and the costs.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of acute pancreatitis，both mild type and severe type

Exclusion Criteria:

* pregnant or suckling
* cancer in late time
* patient near death

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-10 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
the time of first defecation | ten days

SECONDARY OUTCOMES:
the time of bowel sounds getting back to normal | ten days

OTHER OUTCOMES:
Hospitalization cost | ten days

CONTACTS AND LOCATIONS:
Overall Officials: Bin Miao, PHD, Study Chair — Beijing Friendship Hospital; Hong Wang, Graduate, Study Director — Beijing Friendship Hospital; Shuwen Zhang, bachelor, Study Director — Beijing Friendship Hospital; Chao Wang, PHD, Principal Investigator — Beijing Friendship Hospital; Yanli Su, PHD, Principal Investigator — Beijing Friendship Hospital; Shirong Li, graduate, Principal Investigator — Beijing Friendship Hospital; Fengwu Li, graduate, Principal Investigator — Beijing Friendship Hospital; Dinghua Xu, graduate, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China